CLINICAL TRIAL: NCT04035928
Title: Pilot Study on High Resolution 3D Digital Scanning for Maxillofacial Prosthetics for Feasibility and Efficacy
Brief Title: Digital Design for Maxillofacial Prosthetics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment never initiated, change of staff
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, David Zopf, Assistant Professor of Otorhinolaryngology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00155762
Record Dates: First submitted 2019-07-10; First posted 2019-07-29 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Prosthetic Treatment; Craniofacial Abnormalities; Maxillofacial Abnormalities
Keywords: prosthetic treatment; rhinectomy
MeSH Terms: conditions — Craniofacial Abnormalities; Maxillofacial Abnormalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D digital scanning for maxillofacial prosthetics (Experimental)
  Interventions: Device: 3D digital scanning for maxillofacial prosthetics

INTERVENTIONS:
Device: 3D digital scanning for maxillofacial prosthetics — The non-invasive Artec Space Spider 3D scanner will be used to image the indicated areas of the patients head and face. In the case of an intraoral defect, the noninvasive TRIOS intraoral 3D scanner will be used. The study may also use nasometry or nasal endoscopy to measure the amount of airflow through the patient's fistula to help guide the design. The software that will be used will create a 3D image of the prosthesis during the patient's clinic appointment. Once a model of the prosthesis is fully designed and manufactured, the patient will return to clinic for a second appointment which may involve fitting and coloring. A subsequent appointment will involve delivery of a successfully fitted and colored prosthesis that the patient will take home.

SUMMARY:
This study will use a 3D scanner to print a 3D model or mold for each patient's prosthesis. The goal of this study to provide patients with a new, faster method of imaging and creating prostheses that preserves the quality of the current method while reducing time spent by both the patient and providers. Patients that are eligible will have a non-invasive 3D scanner (Artec Space Spider) to image the indicated areas of their head and face to help create their new prosthesis. Patients will come in for visits as needed to fit and adjust their prosthetic. Additionally, patients will be asked to complete questionnaires and have follow-up visits at certain time -points pre and post prosthetic completion.

ELIGIBILITY:
Inclusion Criteria:

* Maxillofacial anatomic defect or anomaly that limits function or cosmesis (including facial and/or intraoral)
* Stable defect (no clinically active tumor or plans for major reconstructive surgery)
* The patient (or family) have elected to pursue a prosthetic reconstruction of a craniofacial anomaly
* The patient is amenable to 3D surface scanning rather than facial molding

Exclusion Criteria:

* Known allergy to silicone
* Poor candidate for prosthetic reconstruction
* Developmental concerns regarding aspiration risk

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Number or weeks to create the final prosthesis | up to 6 months
Time the participants spend in the clinic | up to 6 months
  This includes time spent with participant to design the prosthetic
Number of hours spent to create the prosthetic | up to 6 months
  The number of hours will be calculated by using the design software, scanners, printing, and modifying the mold and prosthesis.

SECONDARY OUTCOMES:
Satisfaction measured by modified Toronto Outcome Measure of Craniofacial Prosthetics (TOMCP) for intraoral prosthesis. | up to 6 months after the prosthetic is completed and being used
  Survey questions are all created using a 7-point Likert scale for assessment. Questions 10-17 from the survey will be used to measure the patients prosthesis level of satisfaction (the higher the score the more satisfied). These will be completed pre-prosthesis and at 1 month and 6 months post prosthesis for patients with intraoral prosthesis.
Satisfaction measured by modified Toronto Outcome Measure of Craniofacial Prosthetics (TOMCP) for extraoral prosthesis. | up to 6 months after the prosthetic is completed and being used
  Survey questions are all created using a 7-point Likert scale for assessment. Questions 8-19 from the survey will be used to measure the patients level of satisfaction (the higher the score the more satisfied). These will be completed pre-prosthesis and at 1 month and 6 months post prosthesis for patients with extraoral prosthesis.
Quality of life measures by modified Toronto Outcome Measure of Craniofacial Prosthetics (TOMCP) for intraoral prosthesis. | up to 6 months after the prosthetic is completed and being used
  Survey questions are all created using a 7-point Likert scale for assessment. Questions 1-9 from the survey will be used to measure the patients level of quality of life (the higher score indicates better quality). These will be completed pre-prosthesis and at 1 month and 6 months post prosthesis for patients with intraoral prosthesis.
Quality of life measures by modified Toronto Outcome Measure of Craniofacial Prosthetics (TOMCP) for extraoral prosthesis. | up to 6 months after the prosthetic is completed and being used
  Survey questions are all created using a 7-point Likert scale for assessment. Questions 1-7 from the survey will be used to measure the patients quality of life (the higher score indicates be better quality). These will be completed pre-prosthesis and at 1 month and 6 months post prosthesis for patients with extraoral prosthesis.
Number of adverse events related to the prosthetic | up to 6 months after the prosthetic is completed and being used
  This study will collect and report adverse events (serious and non-serious) at least possibly related to the prosthetic.

CONTACTS AND LOCATIONS:
Overall Officials: David Zopf, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States